CLINICAL TRIAL: NCT01670591
Title: Effects of Prevention in School (PS): a Swedish School-wide Positive Behavior Support Program at the Primary Prevention Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Bodin, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-12050/2008
Record Dates: First submitted 2012-08-15; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Problem Behaviors Among Students; Classroom Learning Environment
MeSH Terms: interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PS - Prevention in School (Experimental): Teachers learn to use the core program components (defining and teaching school rules and the handling of rule breakings, principles of positive behavior support)with help from external consultants during approximately 1.5 years.
  Interventions: Behavioral: PS - Prevention in School
- Business as usual (No Intervention)

INTERVENTIONS:
Behavioral: PS - Prevention in School
  Arms: PS - Prevention in School

SUMMARY:
Prevention in School (PS) is a modified School-Wide Positive Behavior Support Program at the universal prevention level, developed by Swedish researchers for the school years 4 -9. By defining and teaching school rules to all teachers and students, and by consistently acknowledging students when meeting behavioural expectations, the program aims to reduce problem behaviours in school areas and to improve the classroom learning climate. Against this background, the purpose of this study is to examine whether PS is more effective than schools' ordinary practices in meeting these goals.

ELIGIBILITY:
Inclusion Criteria:

* Schools situated in Stockholm county and in bordering counties within travelling distance from Stockholm.
* Comprising the grades 4-9 (10-15 years).
* A minimum of 2 classes/50 students in each of the grades 5-7.
* A majority (min.80%)of the staff is positive towards program participation.
* School management willing to take active part in change/developmental work.
* A willingness to submit to study conditions (randomization etc)

Exclusion Criteria:

* Participation in other ongoing research projects.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3207 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Student problem behaviors | 24 months
  1. Teacher-reported problem behaviors in school areas during last week
  2. Teacher-reported problem behaviors in classrooms during last week
  3. Student-reported problem behaviors in school areas during the school-year
  4. Student-reported problem behaviors in classrooms during the school-year

SECONDARY OUTCOMES:
Classroom learning climate | 24 months
  1. Teacher self-reports; Teacher Classroom Climate Scale
  2. Student self-reports; Student Classroom Climate Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bodin, Principal Investigator — STAD, Stockholm Centre for Psychiatric Research and Education, Karolinska Institutet
Locations (1):
- STAD, Stockholm Centre for Psychiatric Research and Education, Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Horner RH, Todd AW, Lewis-Palmer T, Irvin LK, Sugai G, & Boland JB. The school-wide evaluation tool (SET): A research instrument for assessing school-wide positive behaviour support. Journal of Positive Behavior Interventions, 6, 3-12, 2004.
- [Background] Sundell K, Koutakis N, Hellqvist A, Andrén J, Karlberg M, Forster M & Hassler-Hallstedt M. Prevention i skolan. Forskningsbaserat preventionsprogram för grundskolans år 4-9. FoU-rapport 2007:6. Stockholms stadsledningskontor: FoU-enheten, 2007.
- [Background] Sørlie M-A, Ogden T. Immediate impacts of PALS: A school wide multi-level programme targeting behaviour problems in elementary school. Scandinavian Journal of Educational Research, 5: 471-492, 2007.
- [Background] Sørlie M-A, Nordahl, T. Problematferd i skolen: Hovedfunn, forklaringer og pedagogiske implikasjoner. [Behaviour problems in school: Main findings, explanations, and pedagogical implications].Hovedrapport fra forskningsprosjektet Skole- och samspillsvansker (Rapport 12a/98). Oslo: Norsk Institutt for forsknings om oppvekst, velferd og aldring, 1998.